CLINICAL TRIAL: NCT00219570
Title: Phase IV Clinical Study Of Clindamycin Phosphate Topical Gel In The Treatment Of Acne Vulgaris
Brief Title: Dalacin-T Gel Post Approval Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Parexel (Industry); SACT INTERNATIONAL Co., LTD. (Unknown); Acronet (Industry); Bellsystem24 , Inc. (Industry); Mitsubishi Kagaku Bio-Clinical Laboratories, inc (Industry); SATO Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A6881003
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; nadifloxacin

INTERVENTIONS:
Drug: clindamycin
Drug: nadifloxacin

SUMMARY:
To investigate, in a comparison vs. Acuatim cream (nadifloxacin cream), the efficacy and safety of Dalacin T Gel (clindamycin phosphate gel) as a therapeutic medication for acne vulgaris in acne vulgaris patients, including children ages 13 and up, in order to clarify the clinical positioning of Dalacin T Gel.

ELIGIBILITY:
Inclusion Criteria:

* Acne vulgaris patients found by a investigator to have at least 10 inflammatory lesions (papules, pustules) on a portion of either a cheeks or the forehead, with an inflammation severity of moderate or worse.

Exclusion Criteria:

* Patients with, for example, acne elastosis, steroidal acne, necrotizing acne, or occupational acne.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2005-01; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To verify the non-inferiority to Acuatim cream of Dalacin T Gel in terms of the percent reduction in the inflammatory lesion count (the assessments of investigator) at Treatment Week 4 or EOT (discontinuation)

SECONDARY OUTCOMES:
To verify the non-inferiority to Acuatim cream of Dalacin T Gel in terms of the percent reduction in the inflammatory lesion count (the assessments of the Data Review Committee based on photographs) at Treatment Week 4 or EOT (discontinuation) According

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer